CLINICAL TRIAL: NCT03070145
Title: Exercise Intervention Among Men With Prostate Cancer Initiating Androgen Deprivation Therapy: A Pilot Study
Brief Title: Exercise Intervention Among Men With Prostate Cancer Initiating Androgen Deprivation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Paul Nguyen, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-515
Record Dates: First submitted 2017-02-06; First posted 2017-03-03 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): * 12-weeks brisk walking and strength training
  * 150 minute moderate aerobic activities, such as brisk walking
  * Strength training 3 days /week
  * One on one sessions with exercise physiologist
  * Optional group sessions
  Interventions: Other: Exercise Intervention
- Usual Care (No Intervention): Usual Care provided

INTERVENTIONS:
Other: Exercise Intervention — 12-week moderate-intensity aerobic and strength training exercise intervention
  Arms: Exercise Intervention

SUMMARY:
This research study is evaluating the impact and feasibility of a 12-week brisk walking and moderate strength training exercise intervention including a virtual component in men who are initiating androgen deprivation therapy (ADT) for prostate cancer

DETAILED DESCRIPTION:
Androgen deprivation therapy (ADT) is a key treatment of prostate cancer. While this therapy improves prostate cancer outcomes, ADT also has a variety of short- and long-term adverse effects, including increased body weight, loss of lean muscle mass, reductions in quality of life, and increased risk of cardiovascular disease. Studies have shown that among men with prostate cancer, physical activity is associated with improved outcomes, including a reduced risk of mortality, from prostate cancer and other causes. Our hypothesis is that physical activity will improve some of the physical and emotional side effects associated with ADT. Physical activity, such as brisk walking and moderate strength training, offers a lifestyle factor that may improve some of the side effects, and is low-cost and easy to do.

The investigators are conducting this study to evaluate the impact and feasibility of a 12-week moderate-intensity aerobic and strength training exercise intervention, including a virtual component. The intervention includes brisk walking and moderate strength training, and involves home-based exercises, in-person sessions with an oncology-trained exercise physiologist, optional group training sessions, and weekly training goals. Participants will have access to a personalized web-based platform called Postwire, which will include videos of training sessions, and will allow participants to easily communicate with the study staff and with other study participants.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any study-related procedures
* History of histologically confirmed prostate cancer
* Initiating or within 30 days of initiating ADT
* ECOG performance status of 0 or 1
* At least 18 years old and no older than 80 years
* Physically able to exercise and have physician consent from their treating physician to start a physical activity program
* English speaking and able to read English
* Have access to and are able to use the internet at a minimum of once per week
* Sufficient proficiency and confidence to use the internet and follow video-based instructions, as determined by the eligibility questionnaire to be completed by the participant
* Willingness to be randomized

Exclusion Criteria:

* Self-reported inability to walk 2 blocks (at any pace)
* Currently physically active (> 90 minutes of moderate or vigorous physical activity per week) as determined by Leisure Score Index of Godin Leisure-Time Exercise Questionnaire [LSI])
* Previously on ADT
* Radiologic evidence of distant disease
* Cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity. Examples would include unstable angina, recent myocardial infarction, oxygen-dependent pulmonary disease, and osteoarthritis requiring imminent joint replacement. Moderate arthritis that does not preclude physical activity is not a reason for ineligibility.
* Psychiatric disorders or conditions that would preclude participation in the study intervention (e.g., untreated major depression or psychosis, substance abuse, severe personality disorder)

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Physical Performance at 12 weeks | Baseline and 12 weeks
  The 6 Minute Walk Test will be performed at the clinic, where the participants will wear tennis shoes and will walk indoors on a flat surface for 6 minutes.
Change from Baseline in Physiologic Measurements at 12 weeks | Baseline and 12 weeks
  Measuring heart rate and resting pulse by counting the number of beats per minute at the wrist of each participant.
Change from Baseline in Blood Pressure at 12 weeks | Baseline and 12 weeks
  The investigators will obtain participant's blood pressure from the most recent clinical visit.
Change from Baseline in Body Composition at 12 weeks | Baseline and 12 weeks
  Obtain body composition (total fat and lean body mass) by conducting dual energy X-ray absorptiometry (DEXA) scans.

SECONDARY OUTCOMES:
Fatigue | Baseline and 12 weeks
  The Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F) is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function.
Physical Functioning | Baseline and 12 weeks
  The investigators will assess changes in physical functioning from study enrollment to the completion of the study period using the European Organization for the Research and Treatment of Cancer (EORTC) QLQ-C30 (version 3) and the Prostate Cancer Specific EORTC questionnaire.
Minutes of Physical Activity | Baseline and 12 weeks
  The investigators will assess changes in activity from baseline to 12-weeks using the 7-Day Physical Activity Recall (PAR)
Anthropometric Measures | Baseline and 12 weeks
  The investigators will assess changes in height from baseline to 12 weeks using a tape measure.
Anthropometric Measures | Baseline and 12 weeks
  The investigators will assess changes in weight from baseline to 12 weeks using a scale.
Anthropometric Measures | Baseline and 12 weeks.
  The investigators will assess changes in waist circumference from baseline to 12 weeks using a tape measure.
Biomarkers | Baseline and 12 weeks.
  The investigators will assess PSA at baseline and 12-weeks in both the usual care and intervention arm.
Biomarkers | Baseline and 12 weeks.
  The investigators will assess testosterone levels at baseline and 12-weeks in both the usual care and intervention arm.
Measure adherence | Baseline and 12 weeks
  The investigators will evaluate adherence rates to study procedures by using self-report and FitBit
Measure feasibility | Baseline and 12 weeks
  Feasibility measured by number of eligible members of the targeted population
Measure feasibility | Baseline and 12 weeks
  Feasibility measured by recruitment rates
Measure feasibility | Baseline and 12 weeks
  Feasibility measured by refusal rates for participation and randomization
Measure feasibility | Baseline and 12 weeks
  Feasibility measured by level of engagement with Postwire and with other study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Paul L. Nguyen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No